CLINICAL TRIAL: NCT00540657
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase II Study Testing CCX282-B in the Treatment of Celiac Disease
Brief Title: A Phase II Study of CCX282-B in Patients With Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL009_282
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — CCX282-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CCX282-B
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CCX282-B — 250mg capsule, twice daily, 13 weeks
  Arms: 1
Drug: Placebo — Placebo capsule, twice daily, 13 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether CCX282-B is effective in mitigating the effects of gluten ingestion in patients with celiac disease

DETAILED DESCRIPTION:
Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, between 18 and 75 years of age
* Established diagnosis of celiac disease
* Subject has been following a strict gluten-free diet for at least 24 months

Key Exclusion Criteria:

* History of any infection requiring intravenous antibiotics, a serious local infection, systemic infection, or gastrointestinal infection within 12 weeks of randomization
* Use of any immunosuppressants, TNF inhibitors, or natalizumab during the 12 weeks prior to study randomization
* Use of steroids during the 4 weeks prior to study randomization
* Receipt of an experimental treatment for any disease within 4 weeks prior to randomization
* Known IgE-mediated atopy or allergy or anaphylactic reactions to gluten
* The subject suffers from a condition that carries a risk at endoscopy or is on anticoagulant treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of CCX282-B compared to placebo on the villous height/crypt depth ratio of small intestinal biopsy specimens taken from subjects with celiac disease, before and after gluten exposure.

SECONDARY OUTCOMES:
Evaluation of CCX282-B compared to placebo on small intestinal mucosal inflammation before and after gluten exposure
Evaluation of CCX282-B compared to placebo on gluten-induced celiac-type serology before and after gluten exposure
Evaluation of CCX282-B compared to placebo on symptom scores before and after gluten exposure

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Finn-Medi Research Ltd, Outpatient Clinic, Tampere, Finland